CLINICAL TRIAL: NCT01158638
Title: Utilizing Tailored Step-Count Feedback to Enhance Physical Activity in the Elderly
Acronym: StepCount
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Scott J. Strath, Associate Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: StepCount; K01AG025962 (NIH)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Physical Activity; Elderly
Keywords: Physical Activity Enhancement
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Usual Care
- 10,000 Steps Group (Active Comparator): Each participant randomized to this study arm will receive a pedometer and a generic recommendation to accumulate 10,000 Steps per Day.
  Interventions: Behavioral: Web Mediated Step Intervention
- Web Mediated Step Group (Experimental): Participants randomized to this study arm receive an introduction to the study website. Each person utilizes the website to track their daily physical activity steps. Goals are given on a weekly basis to increase steps by 10% per day per week over baseline values. The website channels each participant through a series of motivational messages designed to increase compliance with recommended physical activity targets
  Interventions: Behavioral: Web Mediated Step Intervention

INTERVENTIONS:
Behavioral: Web Mediated Step Intervention — The testing of a web mediated step intervention designed to set weekly step targets, and channel participants through a series of motivational screens depending on compliance or non-compliance with set step goals.
  Arms: 10,000 Steps Group; Web Mediated Step Group

SUMMARY:
Individually tailored, mediated pedometer feedback will provide an effective method to promote physical activity adoption in the elderly

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals living in the community.
2. Aged between 50 and 85 years, at screening.
3. Sufficient physical function not to have limitations to participate in physical activity demonstrated by:

   * Habitual gait speed ≥ 1.5 mph, AND
   * No use of a cane or walker, AND
   * Able to walk ≥ 50 feet unaided
4. Sufficient cognitive function, as demonstrated by responses to the mini-mental state examination(>23 score).
5. Be able to read and write in English
6. Sedentary behavior, demonstrated by no regular activity / exercise for previous 6 months and/or a Stage of Change 2 and 3

Exclusion Criteria:

1. Presence of a rapidly progressive or terminal illness condition that is expected to result in significant functional decline during the course of the proposed studies.
2. Significant uncontrolled cardiovascular disease and conditions, e.g. unstable or new onset angina, unrepaired aortic aneurysms, critical aortic stenosis or CAD without bypass, persistent moderate to severe uncontrolled hypertension.
3. Significant uncontrolled metabolic disease, e.g. hemoglobin A1c levels greater than 8.0 and/or glucose levels greater than 300 mg/dL.
4. Fracture of lower extremity within three months.
5. Amputation other than toes.
6. Current history of severe arthritis or orthopedic condition precluding physical activity.
7. Participation in any regular structured exercise (resistance training, Tai Chi, high intensity walking, jogging, cycling, stair climbing, stepping, within the previous 6 months.
8. Individuals that start a new medication that can impact health variables examined during study period (e.g., beta blockers, glucose or cholesterol altering medications), or individuals who alter medication dose that can impact health variables examined within study period.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Objectively assessed steps per day | 12 weeks
  Pedometer determined physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Strath, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- Physical Activity & Health Research Laboratory, Milwaukee, Wisconsin, United States